CLINICAL TRIAL: NCT00923195
Title: Phase II Study of Metastatic Melanoma Using a Chemoradiation Lymphodepleting Conditioning Regimen Followed by Infusion of Anti-Mart-1 and Anti-gp100 TCR-Gene Engineered Lymphocytes and Peptide Vaccines
Brief Title: Radiation, Chemotherapy, Vaccine and Anti-MART-1 and Anti-gp100 Cells for Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090051; 09-C-0051; NCT00814684 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Melanoma; Skin Cancer
Keywords: Metastatic Melanoma; Tumor Regression; Safety; Immunotherapy
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Peptides; montanide ISA 51; Radiation; aldesleukin; Interleukin-2; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TBI 600cGy + PBL + HD IL-2+gp100:154-162 (Experimental): Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population). One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14. Within 24 hours of cell infusion administration of aldesleukin will be initiated as 720,000 IU/kg/dose IV over 15 minutes every 8 hours for up to 5 days (maximum 15 doses).Radiation: 2Gy of TBI twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute.
  Interventions: Drug: Montanide ISA 51 VG; Drug: gp100:154-162 Peptide; Procedure: Radiation; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Genetic: Anti-gp 100:154 TCR PBL
- TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L) (Experimental): Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population). One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14. Within 24 hours of cell infusion administration of aldesleukin will be initiated as 720,000 IU/kg/dose IV over 15 minutes every 8 hours for up to 5 days (maximum 15 doses).Radiation: 2Gy of TBI twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute.
  Interventions: Drug: MART-1: 26-35(27L) Peptide; Drug: Montanide ISA 51 VG; Procedure: Radiation; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Genetic: Anti-MART-1 F5 TCR PBL

INTERVENTIONS:
Drug: MART-1: 26-35(27L) Peptide — Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14.
  Arms: TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)
Drug: Montanide ISA 51 VG — Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14.
Drug: gp100:154-162 Peptide — Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14.
  Arms: TBI 600cGy + PBL + HD IL-2+gp100:154-162
Procedure: Radiation — 2Gy of TBI twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute
Drug: Aldesleukin — Within 24 hours of cell infusion administration of aldesleukin will be initiated as 720,000 IU/kg/dose IV over 15 minutes every 8 hours for up to 5 days (maximum 15 doses).
  Other Names: IL-2; Interleukin-2
Drug: Fludarabine — Day -6 to -2: Fludarabine 25 mg/m2/day IVPB daily over 15-30 minutes for 5 days
  Other Names: Fludara
Drug: Cyclophosphamide — Day -6 to -5: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna15 mg/kg/day over 1 hr X 2 days.
  Other Names: Cytoxan
Genetic: Anti-gp 100:154 TCR PBL — Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or theMART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14
  Arms: TBI 600cGy + PBL + HD IL-2+gp100:154-162
Genetic: Anti-MART-1 F5 TCR PBL — Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or theMART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14
  Arms: TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)

SUMMARY:
Background:

* Melanoma antigen recognized by T-cells (MART-1) and gp100 are two genes found in melanoma cells. An experimental procedure developed for treating patients with advanced melanoma uses these genes and a type of virus to make special cells called anti-MART-1 and anti-gp100 cells, which are designed to destroy the patient's tumor. The cells are created in the laboratory using the patient's own tumor cells or blood cells.
* The procedure also uses one of two vaccines-the anti-MART-1 peptide or the anti-gp100 peptide-to stimulate cells in the immune system that may increase the effectiveness of the anti-MART-1 and anti-gp100 cells. Both vaccines are made from a virus that is modified to carry a copy of the MART-1 gene or gp100 gene. The virus cannot cause disease in humans.

Objectives:

- To evaluate the safety and effectiveness of anti-MART-1 and anti-gp100 cells and peptide vaccines for treating patients with advanced melanoma.

Eligibility:

- Patients 18 years of age with metastatic melanoma for whom standard treatments, including aldesleukin (IL-2) therapy to boost immune response, have not been effective.

Design:

* Participants have an initial evaluation with complete medical history, as well as scans, x-rays, and other tests as directed by researchers. Most of the treatments for this study will be given on an inpatient basis.
* Before the treatment begins, participants will undergo leukapheresis (removal of selected blood cells) to obtain cells for preparing the anti-MART-1 and anti-gp100 cells, and for later stem cell transplantation.
* Preinfusion treatment: 5 days of chemotherapy and 2 days of total-body irradiation to prepare the immune system for receiving the anti-MART-1 and anti-gp100 cells.
* Infusion of cells, followed by IL-2 treatment to improve immune response. IL-2 is given as a 15-minute infusion through a vein every 8 hours for a maximum of 15 doses (over 5 days).
* After the cell infusion, participants will be divided into two groups and will receive either the gp100 peptide or MART-1 vaccine, given once a week for 3 weeks. Participants will also have stem cell transplantation (from previously collected stem cells) to promote cell survival.
* Periodic follow-up clinic visits after hospital discharge for physical examination, review of treatment side effects, laboratory tests and scans every 1 to 6 months.

DETAILED DESCRIPTION:
Background:

* We have engineered human peripheral blood lymphocyte (PBLs) to express a T-cell receptor (TCR) that recognizes human leukocyte antigens (HLAA*0201) restricted epitopes derived from the gp100 or the MART-1 melanoma antigen.
* We constructed single retroviral vectors that contain both Alpha and Beta T cell receptor (TCR) chains and can mediate genetic transfer of this TCR with high efficiency (greater than 30 percent) without the need to perform any selection.
* In co-cultures with HLA-A*0201 positive melanomas these TCR transduced T cells secreted significant amount of interferon-gamma (IFN-y) but no significant secretion was observed in control co-cultures.
* gp100:154-162 TCR or MART-1:27-35 TCR transduced T-cells could efficiently kill HLAA*0201 positive tumors. There was little or no recognition of normal fibroblasts.
* Adoptive transfer of either of these TCR transferred gene modified peripheral blood lymphocyte (PBL) following a nonmyeloablative lymphodepleting regimen could mediate tumor regression in from 13-30 percent of patients with metastatic melanoma though no complete responses were seen.

Objectives:

Primary objectives:

* In cohort 1 and 2, to determine if the administration of both the anti-gp100:154-162 TCR-engineered and anti- MART-1:27-35 TCR-engineered peripheral blood lymphocytes (PBL), aldesleukin and either the gp100:154-162 peptide or the MART-1:26-35(27L) peptide to patients following a chemoradiation lymphodepleting preparative regimen will result in complete tumor regression in patients with metastatic melanoma.
* In cohort 3 and 4, to determine if the administration of both the anti-gp100:154-162 TCR-engineered and anti-MART-1:27-35 TCR-engineered CD8+ peripheral blood lymphocytes (PBL), aldesleukin and either the gp100:154-162 peptide or the MART-1:26-35(27L) peptide to patients following a chemoradiation lymphodepleting preparative regimen will result in complete tumor regression in patients with metastatic melanoma.
* Determine whether the administration of the specific vaccine (the gp100:154-162 peptide or the MART-1:26-35(27L) peptide) can increase the persistence of the specific transferred cells (anti-gp100:154-162 TCR PBL, anti-gp100:154-162 TCR CD8+ PBL, the anti-MART- 1:27-35 TCR PBL, or the anti-MART-1:27-35 TCR CD8+ PBL), respectively.

Secondary objectives:

- Determine the toxicity profile of these treatment regimen.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have:

* metastatic melanoma with measurable disease
* been previously treated with IL-2 for melanoma;
* normal values for basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;
* contraindications for high dose aldesleukin administration.

Design:

* In cohort 1 and 2:

  * Peripheral blood mononuclear cells (PBMC) will be obtained by leukapheresis (approximately 5 times 10(9) cells) and cultured in the presence of anti-CD3 (OKT3) and aldesleukin and separate aliquots will be transduced with the anti-gp100:154-162 TCR and the anti-MART-1:27-35 TCR retroviral vector.
  * Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) cells to supernatant containing the retroviral vectors. These gp100 and MART-1 TCR transduced cells will be separately expanded and tested for their anti-tumor activity.
  * Once engineered lymphocytes are demonstrated to be biologically active according to the strict criteria outlined in the Certificate of Analysis, patients will receive a chemoradiation lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine and 600 cGy total body irradiation followed by intravenous infusion of ex vivo tumor reactive, gp100 and MART-1 TCR gene-transduced cells plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses).
  * Patients will be randomized to receive either the gp100:154-162 peptide or the MART-1:26-35(27L) peptide emulsified in incomplete Freund's adjuvant.
  * Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
  * The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled into each of two cohorts. If none of the 21 patients per cohort experiences a complete clinical response, then no further patients will be enrolled but if 1 or more of the first 21 evaluable patients enrolled in that cohort have a complete clinical response, then accrual to that cohort will continue until a total of 41 evaluable patients have been enrolled in that cohort.
  * Cohort 1 and 2 will be closed with the approval of amendment D.
* Cohort 3 and 4 will be initiated with approval of amendment D.

  * Peripheral blood mononuclear cells (PBMC) will be obtained by leukapheresis (approximately 5 times 10(9) cells) and CD8+ cells will be selected from the cultures, using the Miltenyi CliniMACS apparatus, prior to being stimulated and transduced. Separate aliquots of CD8+ cells will be transduced with the anti-gp100:154-162 TCR and the anti-MART-1:27-35 TCR retroviral vectors.
  * Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) CD8+ cells to supernatant containing the retroviral vectors. These gp100 and MART-1 TCR transduced cells will be separately expanded and tested for their anti-tumor activity.
  * Once engineered lymphocytes are demonstrated to be biologically active according to the strict criteria outlined in the Certificate of Analysis, patients will receive a chemoradiation lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine and 600 cGy total body irradiation followed by intravenous infusion of ex vivo tumor reactive, gp100 and MART-1 TCR gene-transduced CD8+ cells plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses).
  * Patients will be randomized to receive either the gp100:154-162 peptide (cohort 3) or the MART-1:26-35(27L) peptide (cohort 4) emulsified in incomplete Freund's adjuvant.
  * Patients will undergo complete evaluation of tumor with physical examination, CT of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
  * The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled into each of cohort 3 and 4. If none of the 21 patients per cohort experiences a complete clinical response, then no further patients will be enrolled but if 1 or more of the first 21 evaluable patients enrolled in that cohort have a complete clinical response, then accrual to that cohort will continue until a total of 41 evaluable patients have been enrolled in that cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic melanoma with measurable disease.
  2. Previously received aldesleukin (IL-2) and have been either non-responders (progressive disease) or have recurred.
  3. Positive for gp100 and melanoma antigen recognized by T-cells (MART-1) (at least 1 plus and greater than 5 percent) as assessed by immunohistochemistry (IHC) in the Clinical Laboratory Improvement Amendments (CLIA) approved test in the Laboratory of Pathology, Center for cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH).
  4. Greater than or equal to 18 years of age.
  5. Willing to sign a durable power of attorney.
  6. Able to understand and sign the Informed Consent Document.
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  8. Life expectancy of greater than three months.
  9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
  10. Must be human leukocyte antigens (HLA-A*0201) positive
  11. Serology:

  <!-- -->

  1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.

  l. Hematology:
  1. Absolute neutrophil count greater than 1000/m^3
  2. White blood cell (WBC) (greater than 3000/mm^3.
  3. Platelet count greater than 100,000/mm^3.
  4. Hemoglobin greater than 8.0 g/dl.

  m. Chemistry
  1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal.
  2. Serum creatinine less than or equal to 1.6 mg/dl.
  3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

  n. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

  o. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

  p. Six weeks must have elapsed since prior anti-CTLA4 (cytotoxic T-lymphocyte antigen 4) antibody therapy to allow antibody levels to decline, and patients who have previously received anti-CTLA4 antibody must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections; coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; myocardial infarction; cardiac arrhythmias; obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Systemic steroid therapy.
5. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
6. History of coronary revascularization
7. Documented left ventricular ejection fraction (LVEF) of less than 45 percent in patients with:

a) Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, 2 degree or 3 degree heart block

b) Age greater than or equal to 60 years old

h. Documented forced expiratory volume 1 (FEV1) less than or equal to 60 percent predicted for patients with:

1. A prolonged history of cigarette smoking (greater than 20 pack/year within the past 2 years)
2. Symptoms of respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Sakaguchi K, Appella E, Yannelli JR, Adema GJ, Miki T, Rosenberg SA. Identification of a human melanoma antigen recognized by tumor-infiltrating lymphocytes associated with in vivo tumor rejection. Proc Natl Acad Sci U S A. 1994 Jul 5;91(14):6458-62. doi: 10.1073/pnas.91.14.6458. PMID 8022805
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Derived] Abate-Daga D, Hanada K, Davis JL, Yang JC, Rosenberg SA, Morgan RA. Expression profiling of TCR-engineered T cells demonstrates overexpression of multiple inhibitory receptors in persisting lymphocytes. Blood. 2013 Aug 22;122(8):1399-410. doi: 10.1182/blood-2013-04-495531. Epub 2013 Jul 16. PMID 23861247

RESULTS

PARTICIPANT FLOW:
Groups:
- TBI 600cGy + PBL + HD IL-2+gp100:154-162; TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L): Day 0:Autologous transduced CD8+PBL (anti-gp100:154 TCR PBL and anti-MART-1 F5 TCR PBL) infusion will be administered intravenously over 20 to 30 minutes (minimum 5 x 10e8 and up to a maximum of 2 x 10e11 of each transduced lymphocyte population).
  One mg of either the gp100:154-162 or the MART-1:26-35(27) emulsified in IFA by deep subcutaneous injection into each thigh to be administered prior to cell infusion and on days 7 and 14 Within 24 hours of cell infusion administration of aldesleukin will be initiated as 720,000 IU/kg/dose IV over 15 minutes every 8 hours for up to 5 days (maximum 15 doses).
  Radiation: 2Gy of TBI twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute
  Day -6 to -2: Fludarabine 25 mg/m2/day IVPB daily over 15-30 minutes for 5 days Day -6 to -5: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna15 mg/kg/day over 1 hr X 2 days.
Period: Overall Study
Arm/Group | TBI 600cGy + PBL + HD IL-2+gp100:154-162 | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBI 600cGy + PBL + HD IL-2+gp100:154-162 | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (4.9) | 47.5 (12.0) | 48.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rates for Patients With Metastatic Melanoma
Description: Complete response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response is a disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression is at least a 20% increase in the sum of the LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD.
Time Frame: Every 4-6 weeks after initial treatment regimen. If the patient has stable disease or tumor shrinkage, complete evaluations will be repeated every 1-3 months.
Measure: Number; unit: Participants
Arm/Group | TBI 600cGy + PBL + HD IL-2+gp100:154-162 | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)
Number analyzed (Participants) | 2 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Progressive Disease | 2 | 2
  Stable Disease | 0 | 0

2. Secondary Outcome: Toxicity Profile
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 32 months
Measure: Number; unit: Participants
Arm/Group | TBI 600cGy + PBL + HD IL-2+gp100:154-162 | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | TBI 600cGy + PBL + HD IL-2+gp100:154-162 | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L)
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 600cGy + PBL + HD IL-2+gp100:154-162 (N=2) | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L) (N=2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 600cGy + PBL + HD IL-2+gp100:154-162 (N=2) | TBI 600cGy+PBL+HD IL-2+MART-1:26-35(27L) (N=2)
Hearing test abnormal (Ear and labyrinth disorders) | 2 (3) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Leukocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 2 (2) | 2 (3)
Sepsis (Infections and infestations) | 1 (1) | 1 (4)
Wound infection (Infections and infestations) | 1 (6) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Low urine output (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter-related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychosis (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No